CLINICAL TRIAL: NCT00776074
Title: 3 Months, Open-Label, Parallel-Group Study of the Pharmacodynamics, Pharmacokinetics and Safety of TAP-144SR 1-month Depot Gelatin-Free vs. Gelatin-Containing Formulation in Female Patients With Uterine Fibroids
Brief Title: A Pharmacodynamic Study of Leuprorelin Gelatin-Free Formulation in Female Subjects With Uterine Fibroids.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Medical Director, Takeda Pharma Gmbh, Aachen (Germany)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENG K001 GF; 2005-005641-19 (EudraCT Number); EC 406 (Other: Takeda ID); U1111-1114-2217 (Registry Identifier: WHO)
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Uterine Fibroids
Keywords: Leiomyoma; Uterine Fibroids; Drug Therapy; Uterine Neoplasms; Fibroid Tumor
MeSH Terms: conditions — Leiomyoma; Uterine Neoplasms | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Leuprorelin (GF) (Experimental)
  Interventions: Drug: Leuprorelin (GF)
- Leuprorelin (GC) (Experimental)
  Interventions: Drug: Leuprorelin (GC)

INTERVENTIONS:
Drug: Leuprorelin (GF) — Leuprorelin (GF) 3.75 mg injection, subcutaneously, once every 4 weeks for up to 12 weeks.
  Other Names: Leuplin; Enantone; Trenantone; TAP-144SR
  Arms: Leuprorelin (GF)
Drug: Leuprorelin (GC) — Leuprorelin (GC) 3.75 mg injection, subcutaneously, once every 4 weeks for up to 12 weeks.
  Other Names: Leuplin; Enantone; Trenantone; TAP-144SR
  Arms: Leuprorelin (GC)

SUMMARY:
The purpose of this study is to determine the pharmacodynamics of leuprorelin gelatin free formulation (GF) to leuprorelin gelatin containing formulation (GC) in female subjects with uterine fibroids.

DETAILED DESCRIPTION:
Gonadotropin-releasing hormone, also called luteinizing hormone releasing hormone, is a neuropeptide hormone released from the hypothalamus. Gonadotropin-releasing hormone binds to specific gonadotropin-releasing hormone receptors in the cell membrane of pituitary gland cells, inducing the cells to produce and release the gonadotropins: luteinizing hormone and follicle-stimulating hormone. Luteinizing hormone and follicle-stimulating hormone are released into the general circulation and stimulate the gonads to produce and release the sex steroids: testosterone and estrogen. Follicle-stimulating hormone also controls gametogenesis.

Suppression of gonadotropin secretion is an effective treatment for conditions such as prostate cancer, endometriosis and central precocious puberty, because these conditions respond to manipulation of the sex steroids. Suppression of gonadotropin secretion can be achieved by administration of gonadotropin-releasing hormone agonists that, after an initial transient stimulation of gonadotropin release, reversibly desensitize pituitary gonadotropin-releasing hormone receptors. Desensitization is thought to occur by down-regulation of the numbers of gonadotropin-releasing hormone receptors and uncoupling of the receptors from the biochemical pathway that leads to gonadotropin release. Termination of gonadotropin-releasing hormone agonist administration reverses the desensitization, and gonadotropin and sex hormone levels return to normal.

There are several marketed gonadotropin-releasing hormone agonists, one of which is TAP-144 (leuprorelin), an active synthetic nonapeptide gonadotropin-releasing hormone analogue. In the present study, the existing leuprorelin 1- month sustained release formulation will be compared with a new gelatin-free 1-month sustained release formulation.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with measurable uterine fibroids confirmed by vaginal or abdominal ultrasound, deemed otherwise healthy.
* A body mass index in the range 18 to 28.
* Oestradiol, progesterone, luteinizing hormone and follicle stimulating hormone results within the range of normal ovarian function.
* Regular menstruation (except for symptoms of fibroids).
* Females of childbearing potential who are sexually active must agree to use barrier contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.

Exclusion Criteria:

* Acute pelvioperitonitis, ovarian cysts, persistent corpus luteum.
* History of bilateral oophorectomy, hysterectomy, or hypophysectomy.
* Clinically relevant abnormal history, physical findings, or laboratory values at the pre-study screening assessment that could interfere with the objectives of the study or the safety of the patient.
* Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the patient participation in the study or make it unnecessarily hazardous.
* Impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease, or history of any psychotic mental illness.
* Presence or history of severe adverse reaction to any drug.
* Participation in other clinical studies of a new chemical entity or a prescription medicine within the previous 3 months.
* Presence or history of drug or alcohol abuse, or smoking of more than 10 cigarettes daily.
* Evidence of drug abuse on urine testing.
* Positive test for hepatitis B, hepatitis C, human immune deficiency virus 1 or human immune deficiency virus 2.
* Severe bleedings from fibroids.
* Anemia (hemoglobin less than 11 g/dL), loss of more than 400 mL blood during the 3 months before the study.
* Use of oral contraceptives or other estrogen containing medication, progestins, danazol, progesterone antagonists, antiandrogens, steroids or gonadotropins which might affect sex steroid production or activity or assay (e.g. norethindrone) within 30 days prior to study enrolment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Percentage of measured E2 (17β-estradiol) Serum Concentrations less than or equal to 30 pg/mL. | Weeks 5 through Final Visit.

SECONDARY OUTCOMES:
Time course of E2 (17β-estradiol) Serum Concentration levels. | At all Visits.
Time course of E2 (17β-estradiol) Serum Concentrations less than or equal to 30 pg/mL. | Week 5 through Final Visit.
Rate of E2 (17β-estradiol) Serum Concentration levels less than or equal to 50, 40 and 30 ng/dL. | At all Visits.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda Pharma Gmbh, Aachen (Germany)